## PHASE I/II STUDY OF IMMUNIZATION WITH DENDRITIC CELLS LOADED WITH TUMOR EXTRACTS IN PATIENTS WITH ADVANCED MELANOMA.

| 1, | |
|---|---|
| explained to and have accepted an exper disease. I understand that this treatment in the extraction of 500 ml of blood, which are cells using biological factors. Subsequent | declare that I am oma of the skin in stage III/IV. I have been imental treatment with the aim of curing my volves taking cells from my own body through then cultured to mature into activated dendritic ly, these cells are mixed with melanoma cell to stimulate an immune response against the |
| I have been informed of the results obtained in patients treated in a similar manner in other countries. I have been explained that I may not necessarily achieve a complete cure and that this outcome is only expected in a proportion of treated patients. I understand that the administration of these vaccines may be accompanied by some adverse effects such as mild fever, induration at the vaccination site, and, in some cases, areas of skin depigmentation. I comprehend that all information derived from this study will be kept confidential and anonymous and that my participation in this research is entirely voluntary. I may withdraw from this treatment at any time of my own free will, without it affecting my regular treatment plan. | |
| Patient's Signature | |
| Dr. Carlos Ferrada Valenzuela<br>MD. Oncologist | Dr. Mercedes López Nitsche<br>MD. Immunologist |



UNIVERSIDAD DE CHILE FACULTAD DE MEDICINA COMITE DE ETICA PARA INVESTIGACION EN SERES HUMANOS

2 9 ENE. 2002

30,

6

## CERTIFICADO DE APROBACION

El Comité de Etica para la Investigación en Seres Humanos de la Facultad de Medicina de la Universidad de Chile certifica haber estudiado los antecedentes del proyecto ESTUDIO FASE I/II DE INMUNIZACION CON CELULAS DENDRITICAS PULSADAS CON EXTRACTOS TUMORALES, EN PACIENTES CON MELANOMA AVANZASO cuyo Investigador Responsable es el Dr. FLAVIO SALAZAR del Programa de Inmunología del Instituto de Ciencias Biomédicas de esta Facultad.

La Comisión no encontró objeciones éticas y le otorgó su aprobación.

DR JUAN PABLO BECA I.
Presidente

JPEI/mis 2001/32